CLINICAL TRIAL: NCT02948231
Title: MERIT Study - Mistral Percutaneous Mitral Valve Repair FIM Study
Acronym: MERIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitralix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-133
Record Dates: First submitted 2016-06-21; First posted 2016-10-28 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mistral (Experimental)
  Interventions: Device: Mistral implantation

INTERVENTIONS:
Device: Mistral implantation — Mistral Implant is implanted in the Mitral valve

SUMMARY:
The Mistral is an investigational device intended for percutaneous trans-catheter repair in high risk for surgery individuals suffering from functional Mitral Regurgitation.

The device system is to be used only in accordance with the approved Investigational Plan on subjects who have signed an informed consent form. Device use is limited to the approved study investigators.

DETAILED DESCRIPTION:
The study is designed to clinically demonstrate device acute safety (Primary Endpoint) along with longer FU device safety and effectiveness evaluation (Secondary Endpoint).

The main objectives of the study are :

* Evaluate the Acute safety of the implanted Mistral device post procedure and at 30 day follow up period.
* Evaluate the long term Safety of the device (3 and 6 months follow up).
* Demonstrate effectiveness of the Mistral device in improving MR.

Primary endpoints:

• Safety: Acute safety. Rate of device related SAE including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event. At discharge and 30 days.

Secondary endpoints:

* • Safety: Safety at 3 and 6 months. Rate of SAEs and device related SAEs at 3, 6 and 12months.
* Effectiveness: MR reduction post-procedure, at discharge and 30 days, 3 and 6 and 12 months. Improved NYHA class and 6MWT distance at 30 days, 3 and 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to comply with all required follow-up evaluations
* Genders eligible for the study: Both genders
* Subject has functional MR of grade 3+ or more
* Subject has left ventricular ejection fraction (LVEF) >20 % and < 40%.
* No contraindications to trans-septal puncture
* Subject is of functional class 3 or more (NYHA)
* The subject is high risk to undergo MV surgery.
* Subject is excluded from other standard of care procedures as determined by center heart team.
* Patients with femoral veins enabling catheterization with 12Fr catheters
* Life expectancy ≥ 1 year

Exclusion Criteria:

* Mitral Stenosis ≥ moderate
* Aortic Stenosis/Insufficiency > moderate
* Subvalvular calcification or calcification of the chordae.
* Subject has a prosthesis valve in the mitral position
* Transcatheter aortic valve replacement (TAVR) within 30 days prior to subject registration
* Subject has a history of a cerebral vascular accident (CVA) or transient ischemic attack (TIA) within the past 3 months.
* Subject has a history of a myocardial infarction (MI) in the past 3 months
* Subject refuses blood transfusion or surgical valve replacement.
* Subject has had a percutaneous interventional or other invasive cardiac or peripheral procedure ≤ 7 days of the index procedure
* Subject has a history of, or has active endocarditis
* Subject has echocardiographic evidence of intra-cardiac mass, thrombus, vegetation or soft-mobile deposits
* Subject is in acute pulmonary edema.
* Subject has hemodynamic instability requiring inotropic or mechanical support.
* Subject has a known hypersensitivity or contraindication to anticoagulant or antiplatelet medication
* Subject has renal insufficiency as evidenced by a serum Creatinine > 3.0mg/dL.
* Subject has ongoing infection or sepsis
* Subject has blood dyscrasias (leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy)
* Subject has an active peptic ulcer or has had gastrointestinal (GI) bleeding within the past 3 months prior to the index procedure
* Subject requires emergency surgery for any reason
* Subject has a known allergy to Nitinol alloys, 316L\304 stainless steel.
* Pregnant or lactating women.
* Patients being dependent upon the sponsor or upon the investigator or upon the investigational site.
* Subject has a known contrast media allergy
* Presence of high degree atrio-ventricular block (2nd or 3rd degree A-V block), or the presence of tri-fascicular block
* According to investigator on site the patient is suffering from a severe end stage disease (e.g. malignancy, severe pulmonary disease, liver disease, renal failure) and has a life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-25 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Safety: Acute safety. Rate of device related SAE including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event. | Until hospital discharge - up to 5 days post procedure day
Safety: Acute safety. Rate of device related SAE including device related mortality, stroke, MI, cardiac tamponade, surgery for failed percutaneous repair and non-elective cardiovascular surgery to treat an adverse event. | at 30 days post-procedure

SECONDARY OUTCOMES:
Safety: Rate of device related SAE | at 3 months post procedure
Safety: Rate of device related SAE | at 6 months post procedure
Safety: Rate of device related SAE | at 12 months post procedure
Effectiveness: MR Grade reduction. | Post procedure (1 hour after implant device has been implanted)
Effectiveness: MR Grade reduction. | Until hospital discharge - up to 5 days post procedure day
Effectiveness: MR Grade reduction. | at 30 days post procedure
Effectiveness: MR Grade reduction. | at 3 months post procedure
Effectiveness: MR Grade reduction. | at 6 months post procedure
Effectiveness: MR Grade reduction. | at 12 months post procedure
Effectiveness: NYHA class (categorization of heart failure extent). | Post procedure (1 hour after implant device has been implanted)
Effectiveness: NYHA class (categorization of heart failure extent) | Until hospital discharge - up to 5 days post procedure day
Effectiveness: NYHA class (categorization of heart failure extent) | at 30 days post procedure
Effectiveness: NYHA class (categorization of heart failure extent) | at 3 months post procedure
Effectiveness: NYHA class (categorization of heart failure extent) | at 6 months post procedure
Effectiveness: NYHA class (categorization of heart failure extent) | at 12 months post procedure
Effectiveness: 6MWT distance. | Post procedure (1 hour after implant device has been implanted)
Effectiveness: 6MWT distance. | Until hospital discharge - up to 5 days post procedure day
Effectiveness: 6MWT distance. | at 30 days post procedure
Effectiveness: 6MWT distance. | at 3 months post procedure
Effectiveness: 6MWT distance. | at 6 months post procedure
Effectiveness: 6MWT distance. | at 12 months post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- ZNA Middelheim, Antwerp, Belgium